CLINICAL TRIAL: NCT03352544
Title: Exercise Training in Patients With Severe Mental Illness. The PsychiActive Project
Brief Title: Exercise in Severe Mental Illness. The PsychiActive Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, Javier Bueno-Antequera, Principal Investigator, Universidad Pablo de Olavide
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTS948AFS17
Record Dates: First submitted 2017-11-10; First posted 2017-11-24 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Exercise Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise training for 12 weeks (aerobic and resistance training trice a week).
  Interventions: Behavioral: Exercise
- Usual treatment (No Intervention): Usual treatment during 12 weeks, coinciding with exercise intervention time frame.

INTERVENTIONS:
Behavioral: Exercise — Exercise training for 12 weeks (aerobic and resistance training trice a week)
  Other Names: Exercise training
  Arms: Exercise

SUMMARY:
The purpose of this randomized controlled trial is to study the effects of exercise on body weight, body composition, anthropometric and fasting blood measures, physical fitness, pulmonary function, quality of life, and lifestyle habits in patients with severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe mental illness established by experienced psychiatrists, aged 18 years or older and stabilized on antipsychotic medication during the last month.

Exclusion Criteria:

Patients with clinical instability, co-morbid substance abuse, or evidence of uncontrolled cardiovascular, neuromuscular and endocrine disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Fat mass | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Lean mass | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Waist girth | 12 weeks
  In millimeters. Using a measuring tape (Harpenden Anthropometric Tape; Holtain, Dyfed, UK) placed at the midpoint between the last rib and the iliac crest
Hip girth | 12 weeks
  In millimeters. Using a measuring tape (Harpenden Anthropometric Tape; Holtain, Dyfed, UK) placed atthe maximum width over the greater trochanters
Blood glucose | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast
Blood cholesterol | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast
Blood triglyceride | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast

SECONDARY OUTCOMES:
Lower body strength | 12 weeks
  In number of full stands. Using the 30-second chair stand test
Upper body strength | 12 weeks
  In number of bicep curls. Using the 30-second arm curl test
Aerobic endurance | 12 weeks
  In meters. Using the 6-min walk test
Lower body flexibility | 12 weeks
  In centimeters. Using the chair sit-and-reach test
Upper body flexibility | 12 weeks
  In centimeters. Using the back scratch test
Dynamic balance | 12 weeks
  In seconds. Using the 8-foot up-and-go test
Static balance | 12 weeks
  In seconds. Using the stork balance test
Forced vital capacity | 12 weeks
  In liters. Using spirometry (Spirolab II. Medical International Research, Rome, Italy)
Health status | 12 weeks
  Using the Short Form 36-Item Health Survey questionnaire version 2. Examines eight domains of physical (physical functioning, physical role, body pain, and general health) and mental health status (vitality, social functioning, emotional role, and mental health). The four physical-domains are summarized into a physical component score, and the four mental-domains constitute a mental component score. Scores range from 0 to 100 points, with higher scores indicating better health status.
Quality of life | 12 weeks
  Using the Tolerability and Quality of Life questionnaire. Score range from 8 to 32 points. Higher lower represent a better quality of life.
Psychopathological symptoms | 12 weeks
  Using the Brief Symptom Inventory-18 questionnaire. Score range from 0 to 72 points. Higher values represent a higher psychopathological severity.
Anxiety symptoms | 12 weeks
  Using the Beck Anxiety Inventory questionnaire. Score range from 0 to 63 points. Higher values represent a higher level of anxiety.
Depression symptoms | 12 weeks
  Using the Beck depression inventory-II questionnaire. Score range from 0 to 63 points. Higher values represent a higher level of depression.
Self-Esteem | 12 weeks
  Using the Rosenberg Self-Esteem Scale. Score range from 10 to 40 points. Higher values represent a higher self-esteem.
Physical activity | 12 weeks
  Using the Short form International Physical Activity Questionnaire. In metabolic equivalent minutes per week. Higher values represent a higher level of physical activity.
Smoking | 12 weeks
  Using the Fagerström nicotine dependence questionnaire. Score range from 0 to 10 points. Higher values represent a higher nicotine dependece.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pablo de Olavide, Seville, Spain